CLINICAL TRIAL: NCT02252991
Title: APACAN study_Adaptated Physical Activity in Cancerology
Brief Title: Adaptated Physical Activity in Cancerology
Acronym: APACAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to include patients
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014-A00091-46
Record Dates: First submitted 2014-09-11; First posted 2014-09-30 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Fatigue; Physical activity
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A with physical activity during the treatment (Other): In the arm A, patients will realise physical activity during the treatment. Blood samples will be realised. Questionnaries will be given to the patients.
  Interventions: Other: physical activity
- Arm B with physical activity after the treatment (Other): In the arm B, the physical activity will be realised after treatment. Blood samples will be realised. Questionnaries will be given to the patients.
  Interventions: Other: physical activity

INTERVENTIONS:
Other: physical activity — Patients will realise physical activity either during their treatment, either after their treatment. They will have practise a physical activity three times per week.

SUMMARY:
This trial will measure the fatigue in breast cancer patients.

Two groups of patients will be realised:

* Arm A: Physical activity during treatment
* Arm B: No physical activity during treatment but after

The aim of the study is to decrease fatigue, with adequate physical activity, in primary breast cancer patients who receive a treatment for their pathology.

DETAILED DESCRIPTION:
This is an open monocentric study, randomized in two parallel arms with a waiting list.

The duration of the physical activty will vary according to the duration of the treatment: from 2 to 6 months.

Several questionnaries (fatigue, quality of life, ...) will be given to patients at the inclusion, at the end of the period of treatment and 3 to 6 months after the end of treatment.

One hundred patients are necessary in this study (fifty in each arm). We expect to a stability of the fatigue in Arm A compared to an increase of the fatigue in arm B.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 75 years (included)
* Patient with a breast tumor, regardless of the stage and size (except metastatic patients)
* Patient with a local recurrence of breast cancer
* Patient with a second non-metastatic breast cancer
* Breast cancer treated, regardless of the surgery, at least by radiotherapy, chemotherapy (neoadjuvant or adjuvant) +/- targeted therapy
* A mandatory social security affiliation.
* Obtaining informed consent in writing, signed and dated.
* Medical certificate of fitness to practice physical (issued by the medical oncologist)

Exclusion Criteria:

* Cancer other than breast cancer and / or associated with breast cancer
* Metastatic Cancer
* in case of surgery before treatment, delay before beginning treatment inferior to 1 month post-surgery
* Men
* Woman pregnant
* Patient with cognitive or psychiatric disorders
* Patients suffering from disability
* Significant alterations in nutritional status (malnutrition with BMI <19, obese with BMI> 40, BMI)
* Cardiac contraindication to physical activity
* Knowledge and understanding of the French language enough not to learn the correct way of self-administered questionnaires or respond to questioning
* Participation in another clinical study with a similar objective
* Inability to reach the centers where physical activity takes place

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Difference between the questionnaries scores MFI 20 (specific fatigue) between baseline and end of treatment. | up to 6 months
  The scores of fatigue at the end of treatment and at the inclusion will be compared.

SECONDARY OUTCOMES:
QLQ-C30 | up to 6 months
  Comparison of the scores of QLQ-C30 assessed at the end of the treatment and at the inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Jean Bignon, MD,PhD, Principal Investigator — Centre Jean Perrin